CLINICAL TRIAL: NCT02991014
Title: Music-based Intervention for the Reduction of Pain and Stress in Healthy Adults
Brief Title: Music-based Intervention for the Reduction of Pain
Acronym: MINTREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Urs Nater, Prof. Dr., University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MINTREP-UN
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pain Perception; Autonomic Nervous System Functioning
Keywords: music intervention; heart rate variability; frequency modulation; pain perception; cold pressor test (CPT)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- researcher-selected frequency-modulated music (Active Comparator)
  Interventions: Behavioral: researcher-selected frequency-modulated music
- researcher-selected non-modulated music (Placebo Comparator)
  Interventions: Behavioral: researcher-selected non-modulated music
- participant-selected non-modulated music (Experimental)
  Interventions: Behavioral: participant-selected non-modulated music

INTERVENTIONS:
Behavioral: researcher-selected frequency-modulated music — Music pieces have been selected in advance by the researchers. Furthermore, musical frequencies have been artificially modulated.
  Arms: researcher-selected frequency-modulated music
Behavioral: researcher-selected non-modulated music — The same music pieces as in the active comparator arm have been selected in advance by the researchers, but no artificial frequency modulation.
  Arms: researcher-selected non-modulated music
Behavioral: participant-selected non-modulated music — Participants bring their own choice of personally preferred music pieces and listen to them during the intervention sessions. There is no frequency modulation in this condition.
  Arms: participant-selected non-modulated music

SUMMARY:
This study aims to compare the impact of listening to frequency-modulated music vs. non-modulated music (both researcher-selected), and to test whether there are differential effects on pain and stress perception. Further, these two conditions will be compared to a third condition, in which participants will be exposed to self-selected non-modulated music. It is hypothesized that both researcher-selected frequency-modulated music and self-selected non-modulated music result in stronger decreases in stress and pain compared to researcher-selected non-modulated music, while it is expected that there will be no differences in researcher-selected frequency-modulated music and self-selected non-modulated music. The intervention consists of ten sessions of music listening in the course of three consecutive weeks.

DETAILED DESCRIPTION:
This study aims to compare the impact of three different music listening interventions on stress and pain parameters. Participants will be assigned randomly to one of the conditions. In order to avoid expectancy-related effects, participants in both the researcher- and self-selected condition are told that they were allocated randomly to frequency-modulated or non-modulated music. Therefore, subjects are fully blinded with regards to frequency-modulation.

The study design is as follows:

* Baseline measurement: assessment of resting state biological parameters and questionnaires, CPT
* Music listening sessions: ten sessions in three consecutive weeks including:

  1. 60 minutes of music listening
  2. CPT following music listening (sessions 1, 3, 6, 10 only)
  3. Assessments: biological and subjective pain and stress parameters; music and mood related parameters
* Post measurement: assessment of resting state biological parameters and questionnaires, CPT
* Follow-up measurement: 4 weeks after intervention, assessment of resting state biological parameters and questionnaires, CPT

Participants respond to health-related questions (chronic stress, stress reactivity, sleep quality, fatigue, menstrual cycle phase) as well as mood and music-related questions at baseline, post-intervention, and follow-up which are assessed as potential outcome, moderator, and/or control variables. In addition, pain and stress parameters (both biological and subjective) are being assessed at baseline, post-intervention and follow-up as well as in the course of the ten music listening sessions. Furthermore, participants respond to specific music and mood related items following each music listening session (e.g. perceived valence, arousal, familiarity, liking, induced emotions, etc.).

It is hypothesized that listening to researcher-selected frequency-modulated music and self-selected non-modulated music results in stronger increases in pain tolerance and stronger decreases in pain intensity from baseline to post compared to listening to researcher-selected non-modulated music. Furthermore, stronger decreases in stress parameters (e.g. increases in HRV) from baseline to post are expected in the researcher-selected frequency-modulated music and self-selected non-modulated music than in the researcher-selected non-modulated music listening condition. Moreover, it is expected that there will be no differences in researcher-selected frequency-modulated music and self-selected non-modulated music with regards to pain and stress parameters. Additionally, it will be tested whether changes in pain parameters are being mediated* by changes in markers of stress-responsive systems (e.g. heart rate variability indices).

Finally, process analysis over the course of the music listening sessions sessions will be conducted with biological and subjective pain and stress indices as well as music and mood related parameters.

*Although checking for spelling mistakes before submitting the first record, a mistake in wording was discovered only after the release of the record and therefore corrected corresponding to our original hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 35 years
* BMI: 18.5 - 30 kg/m²
* full command of the German language
* capability to attend ten sessions of music listening in our laboratory within three consecutive weeks, each for a duration of one hour

Exclusion Criteria:

* music related profession or studies
* absolute hearing (self-report)
* physical conditions (self-report): tinnitus, hearing impairments, extreme visual impairment, cardiovascular diseases, diabetes, artery occlusive disease, hyper-/hypotension, Raynaud syndrome, chronic pain condition
* pregnancy, breastfeeding
* current mental disorders (self-report): major depression, anxiety disorder, eating disorder, substance dependence, psychosis, schizophrenia
* regular intake of pain drugs/psychotropic drugs
* not being able to refrain from smoking for 2.5 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain Tolerance | Pre-Post-Change-Design: change from baseline to after 3 weeks
  Cold pressor test (CPT): Duration in seconds from immersion of one hand into cold water until removal of the hand:
  * baseline before music intervention
  * post assessment after completion of music intervention (3 weeks)
Pain Intensity | Pre-Post-Change-Design: change from baseline to after 3 weeks
  Cold pressor test (CPT): Subjective pain intensity of the test rated via visual analog scale at the time of removal of the hand
  * baseline assessment before music intervention
  * post assessment after completion of music intervention (3 weeks)

SECONDARY OUTCOMES:
Subjective Stress Experience | Pre-Post-Change-Design: change from baseline to after 3 weeks; process analysis during the course of the intervention
  visual analog scales
  * baseline assessment (before and after CPT)
  * post assessment after completion of music intervention (before and after CPT)
  * in each music listening session (T1: before music listening, T2: after 60 minutes music listening, before CPT; T3: after CPT)
Subjective Stress Experience | Pre-Post-Change-Design: change from baseline to after 3 weeks
  Measurements:
  * chronic stress: SSCS (Screening scale of the TICS - Trier Inventory of Chronic Stress, assessed at baseline and post after completion of music intervention)
  * stress reactivity: PSRS-23 (Perceived Stress Reactivity Scale, assessed at baseline and post after completion of music intervention)
Physiological Stress: Heart Rate Variability Indices | Pre-Post-Change-Design: change from baseline to after 3 weeks, process analysis during the course of the intervention
  Various parameters (e.g. RMSSD, HF, LF, HF/LF)
  * resting state assessed at baseline and post after completion of music intervention
  * continuous assessment in each music listening session
  * assessment in response to CPT
Physiological Stress: Electrodermal activity (EDA) | Pre-Post-Change-Design; change from baseline to after 3 weeks, process analysis during the course of the intervention
  skin conductance level, skin conductance response
  * resting state assessed at baseline and post after completion of music intervention
  * continuous assessment in each music listening session
  * assessment in response to CPT
Physiological Stress: Hair Cortisol | Pre-Post-Change-Design, change from baseline to 4 weeks after post assessment
  Hair Cortisol assessment:
  * baseline before music intervention
  * follow-up assessment 4 weeks after post assessment

OTHER OUTCOMES:
Fatigue | Pre-Post-Change-Design; change from baseline to after 3 weeks
  MFI-20 (Multidimensional Fatigue Inventory)
  * baseline before music intervention
  * post assessment after completion of music intervention (3 weeks)
Sleep Quality | Pre-Follow Up-Change-Design; change from baseline to 4 weeks after post assessment
  PSQI (Pittsburgh Sleep Quality Index)

CONTACTS AND LOCATIONS:
Overall Officials: Urs Nater, PhD, Principal Investigator — University of Vienna
Locations (2):
- University of Vienna, Vienna, Austria
- Philipps-University Marburg, Department of Psychology, Clinical Biopsychology, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feneberg AC, Kappert MB, Maidhof RM, Doering BK, Olbrich D, Nater UM. Efficacy, Treatment Characteristics, and Biopsychological Mechanisms of Music-Listening Interventions in Reducing Pain (MINTREP): Study Protocol of a Three-Armed Pilot Randomized Controlled Trial. Front Psychiatry. 2020 Nov 4;11:518316. doi: 10.3389/fpsyt.2020.518316. eCollection 2020. PMID 33329075